CLINICAL TRIAL: NCT05702177
Title: Single-center, Randomized, Double-blind, Single-dose, 3-way Crossover Study to Compare the Effects of Daridorexant and Placebo on Postural Stability, the Auditory Awakening Threshold, and Cognitive Function in the Middle-of-the-night Following Evening Administration to Healthy Adult and Elderly Subjects
Brief Title: A Study of the Effect of Daridorexant on Nighttime Body Posture, the Noise Level Required to Wake up, and the Ability to Remember Words Previously Presented
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: ID-078-118; 2022-002922-28 (EudraCT Number); NL83038.056.22 (Other: CCMO)
Record Dates: First submitted 2023-01-05; First posted 2023-01-27 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Healthy
MeSH Terms: interventions — daridorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Daridorexant 25 mg (Experimental): Subjects will receive a daridorexant 25 mg tablet for oral administration.
  Interventions: Drug: Daridorexant 25 mg
- Daridorexant 50 mg (Experimental): Subjects will receive a daridorexant 50 mg tablet for oral administration.
  Interventions: Drug: Daridorexant 50 mg
- Placebo (Placebo Comparator): Subjects will receive a daridorexant-matching placebo tablet for oral administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Daridorexant 25 mg — A single-dose of daridorexant 25 mg will be administered in the evening 30 minutes prior to bedtime.
  Other Names: Quviviq
  Arms: Daridorexant 25 mg
Drug: Daridorexant 50 mg — A single-dose of daridorexant 50 mg will be administered in the evening 30 minutes prior to bedtime.
  Other Names: Quviviq
  Arms: Daridorexant 50 mg
Drug: Placebo — A single-dose of placebo matching daridorexant will be administered in the evening 30 minutes prior to bedtime.
  Arms: Placebo

SUMMARY:
A Study of the Effect of Daridorexant on Nighttime Body Posture, the Noise Level Required to Wake up, and the Ability to Remember Words Previously Presented

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in a language understandable to the subject prior to any study-mandated procedure.
* Male and female subjects aged 18 years or older at Screening (18 subjects must be 65 years or older).
* Woman of childbearing potential (WoCBP) who has a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day 1 pre-dose. She must agree to use consistently and correctly (from Screening, during the entire study, and for at least 5-7 days after last study treatment administration) an acceptable method of contraception with a failure rate of less than 1% per year, be sexually inactive, or have a vasectomized partner. If a hormonal contraceptive is used, it must be initiated 1 month before first treatment administration.
* Woman of non-childbearing potential, i.e., postmenopausal (defined as 12 consecutive months with no menses without an alternative medical cause, confirmed by a follicle-stimulating hormone [FSH] test), with previous bilateral salpingectomy, bilateral-oophorectomy or hysterectomy, or with premature ovarian failure (confirmed by a specialist), XY genotype, Turner syndrome, or uterine agenesis.
* Body mass index (BMI) of 18.0 to 35.0 kg/m2 (inclusive) at Screening.
* Ability to communicate well with the investigator, in a language understandable to the subject, and to understand and comply with the study requirements.

Exclusion Criteria:

* Known hypersensitivity to daridorexant, or treatments of the same class, or any of its excipients.
* Any known factor or disease (e.g., unstable medical condition, significant medical disorder, or acute illness) that might interfere with subject's safety, study conduct, or interpretation of the results, such as

  * History of narcolepsy.
  * Shift work within 2 weeks prior to Screening, or planned shift work during the study.
  * Travel across 3 or more time zones within 1 week prior to Screening, or planned travel across 3 or more time zones during the study.
* Previous (i.e., within 2 weeks prior to first study treatment administration) and ongoing treatment with any prescribed central nervous system (CNS)-active medications, and/or diuretics that would affect nighttime rest, and/or moderate to strong cytochromes P450(CYP)3A4 inhibitors or inducers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Treatment difference in postural stability (daridorexant and placebo) | Approximately 4 hours post-dose on Day 2 of the treatment period (daridorexant and placebo). Total duration: 12 hours.
  Postural stability in the MOTN (at 4 h post-dose) evaluated by body sway. Body sway will be assessed approximately 5 min after awakening, with the subject standing comfortably, with eyes closed, using a body sway meter (string attached to the waist). Body movements over 2 min are integrated and expressed as mm sway.

SECONDARY OUTCOMES:
Treatment difference in auditory awakening threshold (daridorexant and placebo) | Approximately 4 hours post-dose on Day 2 of the treatment period (daridorexant and placebo). Total duration: 12 hours.
  The auditory awakening threshold will be assessed at 4 h post dose by applying a 1000 Hz tone, starting at a noise level of 35 dB, increasing in steps of 5 dB until either the subject is awake, or the maximum noise level (100 dB) is reached. The tone will be delivered via a calibrated loudspeaker for 3 s with a 15 s interval between the different noise levels. The subjects must confirm awakening by verbally saying "I'm awake" or similar response, e.g., waving a hand. If a subject does not respond after receiving the initial 100 dB tone, additional 100 dB stimuli will be applied in 15 s intervals for up to 2 min. The outcome measure is the noise level (dB) at which subjects indicate that they are awake. If a subject remains asleep, he/she will be physically awakened by a technician. If a subject will not awaken to any of the tones presented, the maximum 100 dB tone will be recorded as the auditory awakening threshold.
Treatment difference in the timed up and go test (daridorexant and placebo) | Approximately 4 hours post-dose on Day 2 of the treatment period (daridorexant and placebo). Total duration: 12 hours.
Treatment difference in the visual verbal learning test (daridorexant and placebo) | Approximately 4 hours post-dose on Day 2 of the treatment period (daridorexant and placebo). Total duration: 12 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Magliocca M, Koopmans I, Vaillant C, Lemoine V, Zuiker R, Dingemanse J, Muehlan C. Nighttime safety of daridorexant: Evaluation of responsiveness to an external noise stimulus, postural stability, walking, and cognitive function. J Psychopharmacol. 2025 Mar;39(3):223-232. doi: 10.1177/02698811241293997. Epub 2024 Dec 6. PMID 39641404